CLINICAL TRIAL: NCT07272122
Title: Reducing Filth Fly Populations and Transmission of Diarrhoeal Pathogens in Harsh Settings: a Cross-over Trial in South Sudan
Brief Title: Reducing Filth Fly Populations and Transmission of Diarrhoeal Pathogens in Harsh Settings
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Mentor Initiative (Other)
Collaborators: University of Nevada, Las Vegas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: UNLV-2025-203; W911SR2510003 (Other Grant/Funding Number: DoD/USAMRDC)
Record Dates: First submitted 2025-09-24; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Diarrheal Diseases
Keywords: Filth flies; Vector control; Conflict displaced people; Temporary shelter; Cross-over trial
MeSH Terms: interventions — Propoxur; Juvenile Hormones; Diflubenzuron

STUDY DESIGN:
Intervention Model Description: 3-period, 3-group, interventional non-randomised cross-over trial with parallel control
Who Masked: Outcomes Assessor
Masking Description: DSMB committee Trial Steering Committee NB: these committees can request unblinding of data if they have serious concerns regarding adverse event monitoring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention)
- Insecticidal paint treatment of pit latrine wall inner surfaces in refugee camps (Experimental): Inesfly® Carbapaint 10 (Inesfly Corporation, Valencia, Spain) is a water-based polymer coating containing a microencapsulated suspension of 1.0% (w/w) propoxur (carbamate), for slow release to prolong efficacy. Propoxur is a non-repellent active ingredient (AI) and when used on pit latrine walls, flies will land on the surface and receive a lethal insecticidal dose. All eligible pit latrines assigned to this intervention arm will be treated with Inesfly® Carbapaint 10 at the beginning of each 6-month implementation phase; pit latrines with at least 3 standing walls, will be eligible.
  Interventions: Other: Long-lasting insecticidal paint - 1.0% (w/w) propoxur
- Insecticide growth regulator treatment of faeces in pit latrines / open defecation sites (Experimental): All eligible pit latrines (with at least 3 standing walls) assigned to this intervention arm will be treated with Dimilin® GR-2 at 0.5 kg/10m2; granules will be sprinkled onto damp sewage per pit latrine. If waste is desiccated, this intervention will be diluted in water and applied as a spray. This intervention will be re-applied to pit latrines and open defecation sites, every month during each 6-month implementation phase.
  Interventions: Other: Insect growth regulator (IGR) - effervescent granule containing 2% diflubenzuron (20g/kg)

INTERVENTIONS:
Other: Long-lasting insecticidal paint - 1.0% (w/w) propoxur — Inesfly® Carbapaint 10 (Inesfly Corporation, Valencia, Spain) is a water-based polymer coating containing a microencapsulated suspension of 1.0% (w/w) propoxur (carbamate), for slow release to prolong efficacy. Propoxur is a non-repellent active ingredient (AI) and when used on pit latrine walls, flies will land on the surface and receive a lethal insecticidal dose. All eligible pit latrines assigned to this intervention arm will be treated with Inesfly® Carbapaint 10 at the beginning of each 6-month implementation phase; pit latrines with at least 3 standing walls, will be eligible.
  Other Names: Inesfly carbapaint 10
  Arms: Insecticidal paint treatment of pit latrine wall inner surfaces in refugee camps
Other: Insect growth regulator (IGR) - effervescent granule containing 2% diflubenzuron (20g/kg) — This intervention will interrupt filth fly development at the larval / pupal stage, to reduce overall population density. All eligible pit latrines (with at least 3 standing walls) assigned to this intervention arm will be treated with Dimilin® GR-2 at 0.5 kg/10m2; granules will be sprinkled onto damp sewage per pit latrine. If waste is desiccated, this intervention will be diluted in water and applied as a spray. This intervention will be re-applied to pit latrines and open defecation sites, every month during each 6-month implementation phase.
  Other Names: Dimilin® GR-2
  Arms: Insecticide growth regulator treatment of faeces in pit latrines / open defecation sites

SUMMARY:
Objectives The main trial objective is to evaluate the efficacy of insecticidal paint (PAINT) or larvicide (LARV), or both interventions combined, on filth fly density and hence transmission of diarrhoeal diseases.

Primary Objective

• To evaluate the efficacy of PAINT or LARV, or both interventions combined, in reducing the number of cases of all-cause diarrhoea (primary epidemiological endpoint).

Secondary Objectives

* To evaluate the efficacy of PAINT or LARV, or both interventions combined, in reducing filth fly density and species composition at the latrine level (primary entomological endpoint).
* To evaluate the efficacy of PAINT or LARV, or both interventions combined, in reducing filth fly density and species composition at the shelter level (secondary entomological endpoint).

Tertiary Objectives

* To assess the impact of PAINT or LARV, or both interventions combined, on enteric pathogen species composition and density (tertiary entomological endpoint).
* To assess the impact of PAINT or LARV, or both interventions combined, on enteric pathogen antimicrobial resistance (AMR) prevalence (tertiary entomological endpoint).

Trial Design The proposed trial will be a 3-period, 3-group, interventional non-randomized cross-over trial with parallel control (Table 1). The unit of intervention will be an individual refugee camp. Each implementation phase will be 6 months, followed by a 2-month wash-out period.

The trial arms will be:

1. No intervention (control arm)
2. Inesfly® Carbapaint 10 insecticidal paint (intervention arm 1)
3. Dimilin® larvicide (intervention arm 2)

DETAILED DESCRIPTION:
Study Setting This study will take place in Maban County, Upper Nile State, South Sudan, which is home to 4 refugee camps. Many refugees originate from Sudan and others from Ethiopia, Eritrea, and Somalia. The 4 camps host 214,531 refugees (102,857 in Doro, 56,695 in Yusuf Batil, 34,795 in Kaya and 20,184 in Gendrassa), according to UNHCR as of 31 March 2025.

The refugee camps shelters are constructed from a mix of locally sourced materials. Most are temporary shelters made from tarpaulin and plastic sheeting, but some use a mixture of wood, mud, thatch and corrugated iron. The latrines primarily comprise polypropylene sheeting suspended by wooden sticks, with an open roof. They are rudimentary and built to be easily replaceable in case of flooding. Camps are designed with a set ratio of latrines to family shelters.

According to recent District Health Information Systems data, the major causes of death among refugee children arriving to the camps are measles and malnutrition. Malaria remains the leading cause of morbidity and mortality, accounting for 66% of outpatient consultations, 30% of admissions and 50% of deaths. Diarrhoeal diseases affect all refugee age groups but are worse among those under 5s, and attributable to 10% of deaths in this age group.

Age Eligibility Criteria: See "Eligibility"

Arms and Interventions: See "Arms and Interventions" Control arm: no intervention

ITNs are the current standard of care in the refugee camps in Maban County. These are distributed every 2-3 years to protect the population from malaria. ITN coverage is expected to be equitable between intervention and control camps. ITNs will not impact filth flies as they are not hematophagous or nocturnal.

The control arm will not receive a placebo intervention; therefore this will be a non-blinded trial at the implementation level.

Intervention arm 1. Information: Inesfly® Carbapaint 10 (Inesfly Corporation, Valencia, Spain) is a water-based polymer coating containing a microencapsulated suspension of 1.0% (w/w) propoxur (carbamate), for slow release to prolong efficacy. While primarily designed and assed for effectiveness in controlling mosquito and tick populations, Inesfly® Carbapaint 10 was developed to mitigate pyrethroid resistance. Previous iterations of Inesfly® insecticidal paint, combining alpha-cypermethrin, d-allethrin and pyriproxyfen, have shown efficacy against triatomine bugs, sandflies, mosquitoes and tsetse flies. Propoxur is a non-repellent active ingredient (AI) and when used on pit latrine walls, flies will land on the surface and receive a lethal insecticidal dose. This intervention tackles both newly emerged flies from faeces present in the latrines and gravid flies attempting to oviposit; acting on adult flies that are highly likely to be contaminated with microorganisms and spread diarrhoeal diseases. All eligible pit latrines assigned to this intervention arm will be treated with Inesfly® Carbapaint 10 at the beginning of each 6-month implementation phase; pit latrines with at least 3 standing walls, will be eligible. Inesfly® Carbapaint 10 will be applied using brushes or paint rollers at 1L/8m2 on cement, stucco, mud or wood surfaces or 1L/10m2 on painted and metallic surfaces. To wash-out Inesfly® Carbapaint 10, different combinations of warm water and locally available cleaning products (mild soaps or detergents) will be used to clean (scrub, if necessary) pit latrine walls to remove the insecticide formulation. Pit latrine walls will be allowed to air dry and bioefficacy monitoring will be performed using wild-caught filth flies in a random subset of 10 pit latrines which were "washed-out". Modified WHO cone bioassays measuring lethal time to 50% mortality (LT50) will assess fly mortality; no fly mortality following prolonged exposure to pit latrine walls will indicate successful wash-out.

Intervention arm 2: Dimilin® GR-2 larvicide is an effervescent granule containing 2% diflubenzuron (20g/kg), an insect growth regulator (IGR). Diflubenzuron interferes with chitin synthesis resulting in the inhibition of mosquito (Anopheles, Aedes and Culex spp.) or fly (Musca domestica and Stomoxys calcitrans) ecdysis. This intervention will interrupt filth fly development at the larval / pupal stage, to reduce overall population density. All eligible pit latrines (with at least 3 standing walls) assigned to this intervention arm will be treated with Dimilin® GR-2 at 0.5 kg/10m2; granules will be sprinkled onto damp sewage per pit latrine. If waste is desiccated, this intervention will be diluted in water and applied as a spray. This intervention will be re-applied to pit latrines and open defecation sites, every month during each 6-month implementation phase.

To prevent filth fly contamination between camps, Doro and Kaya camps will receive the study interventions since they are more than 7 km apart (29.4 km), based on maximum filth fly dispersal range. Yusuf Batil and Gendrassa (2.6 km apart) will be the parallel control camps throughout the study period; Kaya is 11.6 km away from Yusuf Batil and 13 km from Gendrassa; Doro is 23.4 km from Gendrassa and 25.8 km from Yusuf Batil.

During each implementation phase, project staff will go pit latrine-to-pit latrine to supervise intervention deployment. At the beginning of each wash-out phase, project staff will go pit latrine-to-pit latrine to supervise removal of the PAINT; the residual efficacy of LARV is 1 month, therefore this intervention will dissipate during the 2-month wash-out period.

Explanation for the Choice of Comparators According to the WHO Vector Control Advisory Group (WHO-VCAG), studies should always have a control group from which data collection occurs contemporaneously. Our trial design includes an untreated control arm, which is generally acceptable when compared against an intervention arm, and trial arms are balanced with respect to standards of care. Our study design will not withhold standard of care for any medical treatment or intervention, in alignment with WHO-VCAG guidance.

Criteria for Discontinuing or Modifying Allocated Interventions:

All participation is completely voluntary, and community members can withdraw at any time with impunity. Study staff may terminate subject participation at any time during the trial, as necessary, if a subject no longer meets the inclusion criteria and/or based on adverse event (AE) and/or severe adverse event (SAE) clinical assessment.

Strategies to Improve Adherence to Interventions:

Because trial interventions are implemented at the camp level, not the shelter level, we do not anticipate any issues of participant intervention adherence. The study team will ensure that interventions are deployed at the correct coverage per camp during each implementation phase. Throughout the entomological monitoring, the study team will also perform periodic spot checks that no modifications have been made to pit latrines and intervention re-treatment may be considered, as appropriate.

Relevant Concomitant Care Permitted or Prohibited During the Trial:

Our study design will not withhold standard of care for clinical management or intervention of any medical condition in either trial arm. Camps assigned to either trial arm will continue to receive balanced humanitarian aid and access to healthcare and other medical services.

Outcomes: See "Outcome Measures"

Participant Timeline:

From enrolment to the end of the cross over trial intervention phases.

Sample Size:

Four years of preliminary data were used to calculate sample sizes, targeting a 20% effect size difference from baseline with 80% power and an overall corrected alpha = 0.05 for 2 age cohorts: children 5 years and under and individuals aged 15 and older. The median diarrhoeal proportion across the 4 study camps was used as the baseline proportion in the estimate: 0.18 for children ≤5 years and 0.03 for individuals ≥15 and older. Additionally, the median autocorrelation among years was 0.13 for ≤5 years old and 0.18 for individuals ≥15 years. Using the time-averaged difference method accounting for multiple proportional comparisons among control and intervention arms, assuming a cross-over design across 3 trial periods, an autoregressive covariance structure based on preliminary data, and accounting for 20% loss to follow-up, the study will target a minimum monthly sample size of 342 individuals per camp for ≤5 years old and 1077 individuals per camp for ≥15 years old. To facilitate sampling, both age groups can be recruited from the same shelter, with shelter serving as a random effect in the statistical analysis.

Latrine-level density of filth flies will be estimated using quadrat sampling. Targeting a mean difference in density with an effect size of 0.40, a power of 80%, and an alpha of 0.05, a total of 60 latrines, or 15 latrines per camp, will be targeted for bi-weekly sampling. Shelter-level entomological data will be collected to determine presence/absence of filth flies using passive bait traps. Given that the outcome of interest is surveillance, we follow the recommendations of model simulation studies indicating that a minimum of 20-30 passive sampling devices be used in each location.

Recruitment All participants will be recruited from the 4 refugee camps (Doro, Kaya, Yusuf Batil and Gendrassa) in Maban County, Upper Nile State, South Sudan. Prior to trial commencement, a tiered and iterative approach will be taken to sensitize the communities to project objectives. Letters of introduction will be sent to each camp manager and local community leaders to seek permission to conduct the study. Camp managers, community leaders and local health staff will be invited to sensitization sessions, where the study team will inform them of the project, explain the procedures and timelines and address any questions or concerns. Due to the changing dynamics of this humanitarian emergency, the research team will continually re-assess camp security and accessibility before trial commencement and throughout each implementation phase. Because new issues can arise at any point, project staff will regularly attend camp meetings throughout the baseline year and implementation years to address any problems and to provide updates of study progress.

During trial baseline, project staff will perform a shelter-to-shelter census, where every shelter and pit latrine will be mapped with a Global Positioning System (GPS) and camp members will be informed of the study, procedures and timelines. Recruitment of participants ≤5 years old or ≥15 years old for the post-intervention cohorts will also occur shelter-to-shelter during the baseline census survey. Cohort recruitment per camp will continue until we reach our sample size of 972 enumerated individuals per camp (348 children ≤5 years and 624 individuals ≥15 years); therefore, we anticipate no missing data or issues of initial participant retention. In each subsequent bi-weekly survey, cohort monitoring will occur at a sentinel site per camp, organized by local healthcare workers and project staff. Our sample size calculation for both cohorts assume a 20% loss to follow up across 6 months, with individuals considered "lost-to-follow-up" if they miss at least 3 consecutive visits per implementation period. Because displaced populations can be mobile and the emergency in South Sudan is dynamic, to address issues of participant attrition between project years, each cohort will be re-enrolled at the beginning of each implementation phase. Despite the instability of this setting, we do not anticipate significant participant loss to follow up per monitoring period, since the MENTOR Initiative has conducted several prior clinical trials in these camps, establishing strong local partnerships and a precedent for high study participant retention. Additional eligible individuals will be recruited per cohort, if we encounter greater than anticipated loss to follow up.

Methods: Assignment of Interventions: Allocation and Implementation Because this is an interventional non-randomized cross-over trial design, sequence generation and concealment for participant randomization are not required. Intervention implementation will occur after completion of trial baseline analyses and verification of underlying assumptions of study power. During implementation phase I, Doro camp will receive PAINT and Kaya camp will receive LARV. During implementation phase II, Doro camp will receive LARV and Kaya camp will receive PAINT. During implementation phase III, Doro and Kaya camps will receive both PAINT and LARV. Participants will be recruited to 2 prospective cohorts for monitoring all-cause diarrhoeal case incidence. Camps have been pragmatically allocated to study arms, to minimize intervention contamination from filth fly dispersal range. Study arms will be balanced on the following criteria: diarrhoeal disease case incidence, pit latrine density and filth fly density. Data on these variables per camp will be collected during the baseline cross-sectional survey.

Methods: Assignment of Interventions: Blinding and Emergency Unblinding Due to the obvious nature of the intervention implementation, study participants and project staff will not be blinded to camp allocation. All data analyses will be performed blinded; only 1 study PI will have access to the unblinded camp codes. Blinded data will be shared with the Data Safety and Monitoring Board (DSMB) who can request unblinding, if they have concerns. If an AE may be related to either intervention and non-emergency unblinding is considered, this will follow recommendations outlined in pre-specified standard operating procedures (SOPs). Emergency unblinding will be considered in instances of a suspected, unexpected SAE to either intervention, as judged by site project staff, following recommendations outlined in pre-specified SOPs.

Methods: Data Collection, Management and Analysis Baseline Census At trial baseline, a census questionnaire will be used to collect demographic details on camp residents, including number of people living in each shelter, number of children, participants' ages, family assets (including owning animals within the camp location, as a composite metric for socio-economic status; SES), shelter construction materials, condition and size, distance to nearest health facility, whether cooking is done inside or outside of the shelter, WASH access, distance to nearest pit latrine and latrine type, and distance to nearest domestic waste site. Census data will be used to randomly select eligible individuals for the 2 active monitoring cohorts in each camp and to estimate intervention quantities required. Every shelter, pit latrine and domestic waste disposal site per camp will be mapped with a GPS.

Epidemiological Monitoring To evaluate the effectiveness of PAINT, LARV (IGR) or PAINT + LARV (IGR) in reducing the number of cases of all-cause diarrhoea, epidemiological data will be collected from 2 sources during baseline and each of 3 implementation phases. We will collect information on 1) diarrhoea incidence from local health facilities; and 2) shelter level diarrhoea incidence using bi-weekly surveys. Passive surveillance data on diarrhoeal cases from camp residents will be obtained from the nearby health facilities. Permission will be sought from these facilities during trial baseline, and bi-weekly data will be collected during each 6-month implementation phase.

For shelter-level diarrhoea monitoring, camp residents will be recruited into 2 cohorts to be followed up through each implementation phase. Study participants will be assigned to 1 of 2 cohorts: ≤5 years old, and ≥15 years old, according to the inclusion criteria in Table 2. The rationale for monitoring both age categories is as follows. Most diarrhoeal studies focus on younger age groups as incidence and mortality caused by diarrhoeal illness is much higher in children ≤5 years. This sentinel age category may suffer from increased transmission from poor sanitation and hygiene practices, and young children with worse nutritional status and reduced immunity are more likely to present with illness of greater clinical severity and are therefore more likely to be reported. Monitoring of this high prevalence cohort will allow us to determine if different combinations of interventions can reduce incidence amongst this vulnerable group experiencing multiple modes of diarrhoeal pathogen transmission. We will also collect diarrhoeal incidence data from camp residents that are ≥15 years old. This older cohort is of particular importance as they may be assumed to have improved hygiene practices; therefore, mechanical transmission of diarrhoeal pathogens by flies may be proportionally greater in this age group than amongst younger children. Monitoring of diarrhoeal incidence in this population will also inform how these different vector control interventions can be used to interrupt disease transmission to military servicemen. In most shelters, we will strive to recruit multiple members of the family - 1 participant in the ≤5 years old cohort and at least 1 participant for the ≥15 years old cohort. Normally, this will be the youngest child and a parent or other adult(s) in the household.

Surveys will be completed bi-weekly at a sentinel site per camp, by surveyors trained in obtaining consent and performing accurate data collection in tablet devices using Kobo Toolbox. The bi-weekly questionnaire will contain questions based off the UNICEF questionnaire for active diarrhoeal surveillance. The UNICEF questionnaire uses the WHO definition of diarrhoea (three or more loose or watery stools in a day) while allowing 2 weeks as the recall period: "Has (NAME) had diarrhoea in the last 2 weeks, that is three or more loose or watery stools in a day?". This allows a coverage of reported diarrhoeal cases for the entire month. Visual tools will be incorporated within the questionnaire to establish if the participant is experiencing diarrhoeal illness and to improve accuracy in reporting. For the ≥15 years old cohort, the survey will contain the Bristol Stool Chart, whereas the ≤5 years old cohort will use the Amsterdam Scale. Each of these scales are specifically designed as visual aids for diarrhoea recognition for these age groups. For each shelter included in the study, basic sociodemographic information will also be collected, along with the occurrence of any AEs or SAEs or other related health symptoms, such as fever, headache, or any other illness that has affected the study participant or any other member of the household within the last 2-week period. Study participants will also be asked about intervention perceived effectiveness and other questions pertaining to WASH access and behaviours. A cohort participant (child ≤5 years or person ≥15 years) will be considered "lost-to-follow-up" if they miss at least 3 consecutive visits per implementation period.

Entomology Monitoring in Sentinel Sites Population Density To evaluate the effectiveness of PAINT, LARV (IGR) or PAINT + LARV (IGR) in reducing filth fly density at the shelter and latrine level, we will collect data about fly densities every two weeks throughout each implementation phase. In each of the four camps, 10 sentinel sites will be randomly selected and maintained throughout each 6-month study cycle, for all entomological monitoring activities.

Data will be collected at the latrine level using a Scudder grill. Every two weeks, in each of the 10 monitoring sentinel sites per camp, the project staff will monitor fly ground resting density around three pit latrines (30 latrines per camp). At each latrine, staff will place a Scudder grill on 4 sites close to the latrine, corresponding to the cardinal directions, to reduce any bias in shade and wind directionality; disturbed flies will be allowed 30 seconds to resettle onto the grill, then a photo of the flies will be taken to later morphologically identify fly species, count and establish an approximate density value. The counts will be repeated in similar weather conditions and around the same time of the day.

In each of the 10 sentinel sites per camp, data will also be collected at the shelter level using iCatchi® fly traps (Intellishift (Pty) Ltd). iCatchi ProMax fly traps are designed for commercial and residential use. These traps are 10L containers which hold 3L of a proprietary fly bait, formulated to maximise fly attractiveness to ensure high capture rates. The container design minimizes spillage and allows for easy set up and maintenance, in different environments, including agricultural settings, waste management sites and urban areas. The traps are placed on the ground outdoors and flies enter the large black container through rectangular holes between the bait bowl and larger trap chamber and are unable to exit; they will eventually die from starvation / dehydration. Twice monthly, during each 6-month study implementation phase, one iCatchi ProMax fly trap will be placed in each of the 10 sentinel sites. It will be baited and placed in a fixed outdoor location (<5 m) amongst consenting shelters for a period of two hours. Each of the 10 traps will be collected at the end of the two-hour period, taken to the field entomology laboratory, and the contents be removed carefully emptied for sample extraction, processing, morphological speciation recording, counting, and immediate preservation in a buffer solution in 15ml centrifuge tubes. Samples will be placed directly into field storage at -20oC for future laboratory analysis and sub-studies.

Shelters and pit latrines in each of the entomological sentinel sites will be eligible for inclusion in the entomological monitoring, provided they received the interventions that they were assigned at the beginning of that implementation phase.

Active Ingredient Efficacy Monitoring:

To monitor PAINT residual efficacy, monthly modified WHO cone bioassays measuring LT50 of wild filth flies collected from study camps will be performed in a random subset of 40 treated pit latrines across sentinel sites, per trial arm assigned to this intervention.

To monitor Dimilin residual efficacy, monthly pyramidal emergence traps will be used to sample emergent flies in a random subset of 40 treated pit latrines across sentinel sites, per trial arm assigned to this intervention.

To assess any changes in filth fly insecticide susceptibility following intervention deployment, resistance monitoring will be performed. At baseline and at 3-months post-implementation, in each 6-month implementation phase, wild filth fly populations will be sampled from all 4 camps and exposed to propoxur or diflubenzuron in adult or larval bioassays, respectively.

Propoxur - Adult Fly Testing Adult bioassays will be performed on both susceptible and local wild caught adult flies (by species). There is limited published sectoral experience in fly susceptibility testing for propoxur therefore the study team will conduct and assess three different methods for feasibility at field level and comparability of results.

Feeding Assay:

Wild populations of filth flies will be either aspirated from pit latrine walls or captured when attempting to land on surfaces / food preparations and will be subjected to exposure to serial dilutions of propoxur (e.g. 1000, 100, 10, 1µg AI/ml) diluted in 20% sucrose solution. In each bioassay 10, uniformly sized flies will be introduced into a 157 ml plastic jar containing a dental wick treated with each insecticide concentration (3 replicates per concentration and an untreated control run in parallel). Fly mortality will be scored after 48 hours at 23 ± 2°C, 50% RH and 12L:12D photoperiod. At assessment, flies will be classed as either: (a) unaffected, giving a normal response (making coordinated movements) when gently stimulated by dropping down the containers, or (b) dead or affected, the latter giving an abnormal response to stimulation or showing abnormal movement.

Residual Contact Assay:

The study team will adapt the WHO bottle assay (designed for testing mosquitoes), coating the bottles inside surface with propoxur. A range of test dilutions of propoxur will be made and used to coat separate assay bottles, plus control bottles. Test dilutions will be recorded, and all assay bottles will be clearly labeled. Replicates of 25 adult living flies will be placed into each assay bottle to rest on the interior glass surfaces treated with different dilutions of propoxur, or the control. Assay bottles will be monitored to evaluate knock down and mortality resulting from tarsal contact over a range of time periods.

The study team will coordinate with an external insectary partner to similarly test the same fly species from susceptible colonies for comparison with wild caught adult flies in the study area.

Topical Application Assay:

Replicates (25) of 3- to 5-day old female flies will receive topical application by delivery of a 0.5-l drop of propoxur (in acetone) to the thoracic notum of using a Hand Micro applicator fitted with a Hamilton syringe. Flies will be held in netted cups and provided with 5 cm dental cotton wicks soaked in 15% sugar water and held in a bioassay chamber at 25 C, 12:12 L:D cycle. Mortality will be recorded after 24 h and 48hrs. Propoxur will be tested in a range of up to 5 dilutions. Control groups will receive acetone alone. A minimum of 3 replicates will be conducted.

Feasibility and results of three different assay techniques will be compared, and in partnership with external fly insectary partners, compared with results on susceptible colony flies. Where evident, results will be used to inform ongoing resistance testing in the three phases of the study.

Diflubenzuron - Fly Immature Stage Testing For larval bioassays, wild gravid filth fly populations will be allowed to oviposit onto organic rearing media (created by mixing 1 L of water and 2 L of dry rearing media comprised of 8 parts Purina fly chow, 10 parts pine shavings, and 1 part fish meal). Per bioassay, groups of 20, 3-day old, 2nd instar larvae will be exposed to serial dilutions of diflubenzuron spiked into rearing media (3 replicates will be performed per concentration with an untreated control run in parallel). Larvae will be left on media at 25oC until all larvae have either developed to adults or died; adult flies and pupae will be collected by flotation in a water bath. Larval mortality will be established by subtracting the number of adult flies and non-emerged pupae. Lethal doses (LDs) required to kill 50%, 95% and 99% of the adult and larval filth fly populations will be established at trial baseline and used to monitor changes in insecticide resistance post-intervention.

Laboratory Analysis

A series of sub studies will be conducted on fly samples collected during each 6-month intervention phase, as follows:

Field Laboratory Testing viability of pathogens inside or on flies will be demonstrated through testing freshly trapped field fly samples for Escherichia coli (E. coli). Flies collected from each sampling location will be sub sampled and transported to a nearby field laboratory. Tests will be conducted on pooled (5) fly samples (pooled by morphologically identified species from each of the ten sampling sites. Each pooled fly sample will be crushed and diluted with PBS in separate cryotubes to create dilutions of 10^0 and a 10^(-2) for each fly pool. Each fly soup dilution will be pipetted onto separate preprepared EC plates, and cefotaxime will be plated onto a third plate, then incubated at 35oC for 24 hours, together with labeled negative control plates. E. coli presence, or not, will be carefully recorded and data input into an Excel spreadsheet. Any fly samples that are TNTC for E. coli at the 10^(-2) dilution will be re-tested.

UNLV Laboratory At least 200 fly samples collected through each of the three intervention phases, across the study arms will be assigned for for laboratory testing in UNLV. These will be immediately preserved in buffer solution in 2 ml Eppendorf tubes and then frozen and stored at -20oC in the field laboratory. A replicate of 200 flies sampled for each intervention phase will also be preserved and retained in freezer storage as a contingency sample.

At the end of each intervention phase 200 of the preserved and frozen fly samples collected during that 6-month phase will be transported to UNLV in a cold chain, for fly and pathogen identification during each wash-out period.

The laboratory analysis will include morphological identification of individual flies to species level, performed according to standard dichotomous taxonomic keys. Per trial 6-month period, 200 randomly sampled flies (split equitably across clusters / trial arms) will be selected for molecular analysis. A total of 600 flies will be analysed over the course of the study. Of these, a subset of at least 100 flies will be analysed using a custom a custom TaqMan Array Card (TAC) initially in order to identify the most prevalent pathogens in the samples. Following the completion of TAC analysis on the subset of 100 flies, a further 500 flies will be analysed by quantitative polymerase chain reaction (qPCR) for the most prevalent targets identified by TAC.

Data Management:

Epidemiological and entomological data will be entered into electronic forms on smartphones or tablets installed with Kobo Toolbox. The data will be stored on a secure server located at the MENTOR Initiative in-country office. All data management and analyses will be performed using STATA/SE 17.0 and R.

Data Quality and Control (QC). SOPs for data collection will be developed, and study data collectors will be appropriately trained to ensure rigorous data collection. QC will be conducted by a supervisor who will monitor the performance of the data collectors.

Statistical Methods - Outcomes To assess differences in diarrhoeal incidence by age group (primary epidemiological outcome) among camps in the intervention and control arms across the 3 time periods, a chi-square multiple proportion test based on a weighted sum of squared deviations to compare observed group proportions to the overall proportion for all groups will be utilized. This analysis will provide a means to assess absolute proportional differences; should overall differences be detected, post-hoc Bonferroni-corrected pairwise proportion tests with bootstrapped p-values will be investigated. Additionally, we will model proportions from each sampled shelter as a dependent variable using a general linear beta regression model. The model will utilize several independent predictors, including age group, camp, time, filth fly intervention, etc. to assess their relationship with overall diarrhoeal proportion, hence allowing for simultaneous prediction of disease outcome as a function of multiple measured and potentially modifiable variables. Outcomes comparing changes in proportions of filth fly species, pathogens and AMR markers will be compared between interventions / camps using mixed-effect logistic regression, accounting for clustering effect and adjusted for baseline fly density and pathogen prevalence. Mixed-effects negative binomial regression analysis will be used to estimate density ratios of the effect of each (or combined) intervention on filth fly populations, compared with control camps. Insecticide susceptibility per trial arm will be estimated using generalized linear mixed models (GLMMs), with random effects of dose and test replicate and fixed effects of trial year and arm.

ELIGIBILITY:
Inclusion Criteria:-

* Individuals of either <5 years old or >15 years old all ages
* Slept in camp ≥27 nights during any given month
* Individual is not severely malnourished, sick, anemic (self-reported), has signs of clinical decompensation, and/or has any other chronic co-morbidities (e.g. HIV or cancer)
* No plans for extended travel (>1 month) outside of camp during study
* Resides in an easily accessible dwelling and is present at time of enrolment
* Not participating in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure during the trial
* Provision of informed consent form signed by the parent(s) or guardian (under 5s), able to give informed consent as an adult or able to give informed assent for children >15 years

Exclusion Criteria:

* Child < 1 years old (due to breastfeeding) or aged >5 and < 15 years old
* Slept in camp <27 nights during any given month
* Individual is severely malnourished, sick, anemic, has signs of clinical decompensation, and/or has any other chronic co-morbidities (e.g. HIV or cancer)
* Plans for extended travel (>1 month) outside of camp during study
* Not present at time of enrolment
* Participating or planning to participate in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure during the trial
* No provision of informed consent form signed by the parent(s) or guardian (under 5s), unable to give informed consent as an adult or unable to give informed assent for children >15 years

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5676 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-19 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of insecticidal paint (PAINT) or insect growth regulator (LARV), or both interventions combined, in reducing the number of cases of all-cause diarrhoea (primary epidemiological endpoint). | At trial baseline and then every fortnight during each of three 6-month intervention phases.
  The primary outcome will be all-cause diarrhoeal case incidence in children <5 and individuals >15. A diarrhoeal case is defined by WHO as the passage of 3 or more loose or liquid stools per day (or more frequent passage than is normal for the individual). Epidemiological data will be collected from 2 sources during baseline and each of 3 implementation phases. We will collect information on 1) diarrhoea incidence from local health facilities; and 2) shelter level diarrhoea incidence using bi-weekly surveys. Passive surveillance data on diarrhoeal cases from camp residents will be obtained from the nearby health facilities. Permission will be sought from these facilities during trial baseline, and bi-weekly data will be collected during each 6-month implementation phase.

SECONDARY OUTCOMES:
Filth fly density and species composition | At trial baseline and then every fortnight during each of three 6-month intervention phases.
  To evaluate the efficacy of PAINT or LARV, or both interventions combined, in reducing filth fly density at the latrine level (primary entomological endpoint).
Filth fly species composition - latrine level | At trial baseline and then every fortnight during each of three 6-month intervention phases.
  To evaluate the efficacy of PAINT or LARV, or both interventions combined, in reducing filth fly species composition at the latrine level (primary entomological endpoint).
Filth fly species density - shelter level | At trial baseline and then every fortnight during each of three 6-month intervention phases.
  To evaluate the efficacy of PAINT or LARV, or both interventions combined, in reducing filth fly density at the shelter level (secondary entomological endpoint).
Filth fly species composition - shelter level | At trial baseline and then every fortnight during each of three 6-month intervention phases.
  To evaluate the efficacy of PAINT or LARV, or both interventions combined, in reducing filth fly species composition at the shelter level (secondary entomological endpoint).

OTHER OUTCOMES:
Impact of PAINT or LARV, or both interventions combined, on enteric pathogen density | At trial baseline and then every fortnight during each of three 6-month intervention phases.
  To assess the impact of PAINT or LARV, or both interventions combined, on enteric pathogen species density (tertiary entomological endpoint).
Impact of PAINT or LARV, or both interventions combined, on enteric pathogen species composition | At trial baseline and then every fortnight during each of three 6-month intervention phases.
  To assess the impact of PAINT or LARV, or both interventions combined, on enteric pathogen species composition (tertiary entomological endpoint)
Impact of PAINT or LARV, or both interventions combined, on enteric pathogen antimicrobial prevalence | At trial baseline and then every fortnight during each of three 6-month intervention phases.
  To assess the impact of PAINT or LARV, or both interventions combined, on enteric pathogen antimicrobial resistance (AMR) prevalence (tertiary entomological endpoint).

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Allan, PhD, Principal Investigator — The Mentor Initiative
Locations (1):
- The MENTOR Initiative, Bunj Town, Maban, Bunj, Maban County, South Sudan

IPD SHARING:
Plan to Share IPD: Yes
Summary findings from trial data will be published in peer reviewed publications and their supporting information. All other relevant de-identified participant data are available from the trial PIs upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: IPD will be available upon publication of the main trial manuscript, following trial completion and will be available indefinitely.
Access Criteria: Summary findings from trial IPD will be published in open-access, peer reviewed papers and their supporting information. Following trial completion, IPD will be available indefinitely, upon publication of the main trial manuscript. All other relevant de-identified IPD are available from the trial Principal Investigators upon reasonable request.

REFERENCES:
- [Background] Council for International Organizations of Medical Sciences. International ethical guidelines for biomedical research involving human subjects. Bull Med Ethics. 2002 Oct;(182):17-23. PMID 14983848
- [Background] Capone D, Cumming O, Flemister A, Ilevbare V, Irish SR, Keenum I, Knee J, Nala R, Brown J. Sanitation in urban areas may limit the spread of antimicrobial resistance via flies. PLoS One. 2024 Mar 20;19(3):e0298578. doi: 10.1371/journal.pone.0298578. eCollection 2024. PMID 38507457
- [Background] Capone D, Adriano Z, Cumming O, Irish SR, Knee J, Nala R, Brown J. Urban Onsite Sanitation Upgrades and Synanthropic Flies in Maputo, Mozambique: Effects on Enteric Pathogen Infection Risks. Environ Sci Technol. 2023 Jan 10;57(1):549-560. doi: 10.1021/acs.est.2c06864. Epub 2022 Dec 14. PMID 36516327
- [Background] Hamer GL, Kelly PH, Focks DA, Goldberg TL, Walkers ED. Evaluation of a novel emergence trap to study Culex mosquitoes in urban catch basins. J Am Mosq Control Assoc. 2011 Jun;27(2):142-7. doi: 10.2987/10-6090.1. PMID 21805846
- [Background] Committee, I. R. A., (IRAC Susceptibility Test Methods Series Method No: 026).
- [Background] Amsterdam, U. o. Constipation in infancy and childhood: New insights into pathophysiological aspects and treatment. https://pure.uva.nl/ws/files/1294622/73258_07.pdf (2010).
- [Background] Australia, C. F. o. Faecal Bristol Stool Chart, 2024).
- [Background] Rego R, Watson S, Alam MAU, Abdullah SA, Yunus M, Alam IT, Chowdhury ASMHK, Haider SMA, Faruque A, Khan AI, Hofer T, Gill P, Islam MS, Lilford R. A comparison of traditional diarrhoea measurement methods with microbiological and biochemical indicators: A cross-sectional observational study in the Cox's Bazar displaced persons camp. EClinicalMedicine. 2021 Nov 20;42:101205. doi: 10.1016/j.eclinm.2021.101205. eCollection 2021 Dec. PMID 34849477
- [Background] Jiménez-Valverde, A. Sample size for the evaluation of presence-absence models. Ecological Indicators 114, 106289 (2020).
- [Background] Organization, W. H. How to design vector control efficacy trials: guidance on phase III vector control field trial design provided by the Vector Control Advisory Group. ttps://iris.who.int/bitstream/handle/10665/259688/WHO-HTM-NTD-VEM-2017.03-eng.pdf (2017).
- [Background] Nazni WA, Luke H, Wan Rozita WM, Abdullah AG, Sa'diyah I, Azahari AH, Zamree I, Tan SB, Lee HL, Sofian MA. Determination of the flight range and dispersal of the house fly, Musca domestica (L.) using mark release recapture technique. Trop Biomed. 2005 Jun;22(1):53-61. PMID 16880754
- [Background] Zaki, A. M., Darwish, E. T. E. & Abdella, M. M. H. Bio-efficacy of certain chitin synthesis inhibitors on dipterous flies and mites inhabiting dung of farm animals. Journal of Pest Science 63, 69-73 (1990).
- [Background] Albayyar, E. A. & Qader, R. A. A. A. Effect of Insect Growth Regulators "Dimilin25% wp and Match 50 EC" Against House Fly (Musca domestica) Life Stages (Diptera: Muscidae). Indian Journal of Forensic Medicine & Toxicology 15, 2867-2870 (2021).
- [Background] Chen K, Deguenon JM, Cave G, Denning SS, Reiskind MH, Watson DW, Stewart DA, Gittins D, Zheng Y, Liu X, Mouhamadou CS, Roe RM. New thinking for filth fly control: residual, non-chemical wall spray from volcanic glass. Med Vet Entomol. 2021 Sep;35(3):451-461. doi: 10.1111/mve.12521. Epub 2021 May 3. PMID 33942346
- [Background] Organization, W. H. Guidelines for Testing Mosquito Adulticides for Indoor Residual Spraying and Treatment of Mosquito Nets. (Geneva, Switzerland, 2006).
- [Background] Acapovi-Yao, G. et al. Assessment of the efficiency of insecticide paint and impregnated nets on tsetse populations: preliminary study in forest relics of Abidjan, Côte d'Ivoire. West African Journal of Applied Ecology 22, 17-25 (2014).
- [Background] Mosqueira B, Duchon S, Chandre F, Hougard JM, Carnevale P, Mas-Coma S. Efficacy of an insecticide paint against insecticide-susceptible and resistant mosquitoes - part 1: laboratory evaluation. Malar J. 2010 Nov 25;9:340. doi: 10.1186/1475-2875-9-340. PMID 21108819
- [Background] Mosqueira B, Chabi J, Chandre F, Akogbeto M, Hougard JM, Carnevale P, Mas-Coma S. Efficacy of an insecticide paint against malaria vectors and nuisance in West Africa--part 2: field evaluation. Malar J. 2010 Nov 25;9:341. doi: 10.1186/1475-2875-9-341. PMID 21108820
- [Background] Mosqueira B, Chabi J, Chandre F, Akogbeto M, Hougard JM, Carnevale P, Mas-Coma S. Proposed use of spatial mortality assessments as part of the pesticide evaluation scheme for vector control. Malar J. 2013 Oct 18;12:366. doi: 10.1186/1475-2875-12-366. PMID 24139513
- [Background] Mosqueira B, Soma DD, Namountougou M, Poda S, Diabate A, Ali O, Fournet F, Baldet T, Carnevale P, Dabire RK, Mas-Coma S. Pilot study on the combination of an organophosphate-based insecticide paint and pyrethroid-treated long lasting nets against pyrethroid resistant malaria vectors in Burkina Faso. Acta Trop. 2015 Aug;148:162-9. doi: 10.1016/j.actatropica.2015.04.010. Epub 2015 May 7. PMID 25959771
- [Background] Poda SB, Soma DD, Hien A, Namountougou M, Gnankine O, Diabate A, Fournet F, Baldet T, Mas-Coma S, Mosqueira B, Dabire RK. Targeted application of an organophosphate-based paint applied on windows and doors against Anopheles coluzzii resistant to pyrethroids under real life conditions in Vallee du Kou, Burkina Faso (West Africa). Malar J. 2018 Apr 2;17(1):136. doi: 10.1186/s12936-018-2273-x. PMID 29609597
- [Background] Alim A, Huda MM, Ghosh D, Halleux CM, Almahmud M, Olliaro PL, Matlashewski G, Kroeger A, Aseffa A, Mondal D. Long-Term Efficacy of Insecticidal Wall Painting for Controlling Visceral Leishmaniasis Vectors in Bangladesh. Am J Trop Med Hyg. 2023 Sep 18;109(5):1022-1027. doi: 10.4269/ajtmh.22-0809. Print 2023 Nov 1. PMID 37722667
- [Background] Alarico AG, Romero N, Hernandez L, Catala S, Gorla D. Residual effect of a micro-encapsulated formulation of organophosphates and piriproxifen on the mortality of deltamethrin resistant Triatoma infestans populations in rural houses of the Bolivian Chaco region. Mem Inst Oswaldo Cruz. 2010 Sep;105(6):752-6. doi: 10.1590/s0074-02762010000600004. PMID 20944988
- [Background] Maloney KM, Ancca-Juarez J, Salazar R, Borrini-Mayori K, Niemierko M, Yukich JO, Naquira C, Keating JA, Levy MZ. Comparison of insecticidal paint and deltamethrin against Triatoma infestans (Hemiptera: Reduviidae) feeding and mortality in simulated natural conditions. J Vector Ecol. 2013 Jun;38(1):6-11. doi: 10.1111/j.1948-7134.2013.12003.x. PMID 23701602
- [Background] Alvarez-Hernandez G, Trejo AV, Ratti V, Teglas M, Wallace DI. Modeling of Control Efforts against Rhipicephalus sanguineus, the Vector of Rocky Mountain Spotted Fever in Sonora Mexico. Insects. 2022 Mar 7;13(3):263. doi: 10.3390/insects13030263. PMID 35323561
- [Background] Mahase E. Measles: South Sudan reports 12 000 cases in three months. BMJ. 2024 Mar 28;384:q777. doi: 10.1136/bmj.q777. No abstract available. PMID 38548295
- [Background] Public Health Weekly Reports for MAY 9, P. H. R. W. & 669-96., D. C. 17 Classification, I. F. S. P. South Sudan: acute malnutrition situation for July - September 2023 and projections for October 2023 - March 2024 and April - June 2024, 2024).
- [Background] (UNHCR), U. N. H. C. F. R. Vector and pest control in refugee situations. (1997). 15 Board, A. F. P. M. Filth Flies: Significance and Control in Contingency Operations Technical Guide No. 30 (2011).
- [Background] Onwugamba FC, Mellmann A, Nwaugo VO, Suselbeck B, Schaumburg F. Antimicrobial resistant and enteropathogenic bacteria in 'filth flies': a cross-sectional study from Nigeria. Sci Rep. 2020 Oct 12;10(1):16990. doi: 10.1038/s41598-020-74112-x. PMID 33046808
- [Background] Graczyk TK, Knight R, Gilman RH, Cranfield MR. The role of non-biting flies in the epidemiology of human infectious diseases. Microbes Infect. 2001 Mar;3(3):231-5. doi: 10.1016/s1286-4579(01)01371-5. PMID 11358717
- [Background] Agency, T. U. R. Refugee population in Maban, South Sudan, 31 October 2023, 2023). 11 Hewitt, C. G. Houseflies and how they spread disease. (1912).
- [Background] Riddle MS, Martin GJ, Murray CK, Burgess TH, Connor P, Mancuso JD, Schnaubelt ER, Ballard TP, Fraser J, Tribble DR. Management of Acute Diarrheal Illness During Deployment: A Deployment Health Guideline and Expert Panel Report. Mil Med. 2017 Sep;182(S2):34-52. doi: 10.7205/MILMED-D-17-00077. PMID 28885922
- [Background] Organization, W. H. Diarrhoeal disease (2024).
- [Background] GBD 2021 Diarrhoeal Diseases Collaborators. Global, regional, and national age-sex-specific burden of diarrhoeal diseases, their risk factors, and aetiologies, 1990-2021, for 204 countries and territories: a systematic analysis for the Global Burden of Disease Study 2021. Lancet Infect Dis. 2025 May;25(5):519-536. doi: 10.1016/S1473-3099(24)00691-1. Epub 2024 Dec 18. PMID 39708822
- [Background] GBD 2019 Under-5 Mortality Collaborators. Global, regional, and national progress towards Sustainable Development Goal 3.2 for neonatal and child health: all-cause and cause-specific mortality findings from the Global Burden of Disease Study 2019. Lancet. 2021 Sep 4;398(10303):870-905. doi: 10.1016/S0140-6736(21)01207-1. Epub 2021 Aug 17. PMID 34416195
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884